CLINICAL TRIAL: NCT07043244
Title: The Effect of Virtual Reality-Based Occupational Health and Safety Training on Workplace Accidents and Occupational Health Literacy Among Adolescents in Vocational Education
Acronym: no one
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025/01; 2025-010 (Other Grant/Funding Number: Saglik Bilimleri University)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Occupational Health; Work Accident; Labor
Keywords: Occupational health literacy, occupational accidents, vocational education, and adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality simulation Participants receive virtual reality-based occupational health and safety (Experimental)
  Interventions: Behavioral: virtual reality simulation
- Control Arm: Participants did not receive any occupational health and safety training. (No Intervention)

INTERVENTIONS:
Behavioral: virtual reality simulation — no description, work attempt completed
  Arms: Virtual reality simulation Participants receive virtual reality-based occupational health and safety

SUMMARY:
In Türkiye, Vocational Education Centers (VECs) provide apprenticeship and mastery training as well as vocational course programs under the regulation of the Ministry of National Education. These centers aim to equip learners with practical and theoretical skills aligned with labor market needs. In VECs, students receive theoretical education one to two days per week, while spending four to five days receiving hands-on vocational training at workplaces. As part of this structure, students are insured against occupational accidents and diseases and receive 30% of the minimum wage. Currently, approximately 1.5 million students are enrolled in VECs, with an employment rate of 88%, significantly higher than that of vocational high schools (55%).

The Motor Vehicles Technology field is one of the most populated programs in VECs. Türkiye's rapid advancement in the automotive industry has heightened the demand for a qualified workforce in this area. According to the UN Convention on the Rights of the Child, Türkiye recognizes every person under 18 years as a child. However, the labor force participation rate among children aged 15-17 has risen to 22.1%. These children often work long hours under unfavorable conditions. Reports indicate that children working in automotive technology suffer from musculoskeletal issues, lack tetanus vaccination, and do not utilize personal protective equipment.

Despite Türkiye's ratification of international conventions addressing child labor, the prevalence of child labor and related adverse social and health consequences remain a challenge. Occupational accidents are alarmingly high among child workers. One critical factor in reducing such incidents is improving Occupational Health Literacy (OHL), defined as the capacity of workers to access, understand, and use information and services to make informed decisions regarding workplace health and safety.

This project aims to reduce work-related accidents and improve the OHL levels of child workers in the Motor Vehicles Technology field through a Virtual Reality (VR) simulation-based occupational health and safety education program. VR simulation provides a three-dimensional, interactive learning environment where users can explore and engage with simulated scenarios. VR is particularly suitable for demonstrating hazardous, costly, or complex processes that are difficult to replicate in classroom settings. According to literature, VR-based learning yields better educational outcomes compared to traditional methods, offering cost-effectiveness, efficient space use, and opportunities for self-directed learning.

The proposed program integrates VR simulations designed to present realistic workplace hazards and safety practices. Through immersive interaction, the program seeks to enhance learners' awareness and behavioral competence regarding occupational risks. This intervention, targeting Generation Z youth, aligns with the urgent need for innovative, tech-supported approaches to safeguard children's health in vocational contexts.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 15 to 18 enrolled in the Motor Vehicles Technology program at Sarıyer Atatürk Vocational Education Center, Residing in Istanbul during the data collection period and able to participate in face-to-face interviews, Officially registered for the 2024-2025 academic year, Regularly attending school, Regularly attending work-based training, Have not previously received virtual reality simulation-based occupational health and safety training, Have no physical or mental disabilities, Capable of using mass communication tools, Have parental consent, Willing to voluntarily participate in the study.

Exclusion Criteria:

Having any physical or mental disabilities, Unwilling to participate in the study, Irregular attendance at school or workplace, Students repeating a grade will be excluded from the study.

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Change in occupational health literacy levels | Baseline, 4 weeks, and 8 weeks after the intervention
  Occupational health literacy will be measured using a standardized questionnaire before and after the VR-based occupational health and safety training. Score changes will reflect effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarıyer Atatürk Vocational Education Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy. Only aggregated findings will be published in scientific articles.